CLINICAL TRIAL: NCT04710667
Title: Sports Science Institute
Brief Title: To Explore the Effects of Different Training Periods and Dietary Pattern on the Gut Microbiota, Metabolites and Protein Expression Levels of Strength and Endurance Athletes and to Find Relevant Biological Indicators.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan Sport University (Other)
Responsible Party: Principal Investigator, LinYuChih, Principal Investigator, National Taiwan Sport University
Other Study IDs: IRB-19-039-B1
Record Dates: First submitted 2021-01-12; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Athlete

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The gastrointestinal tract contains hundreds of millions of microorganisms, collectively called the intestinal flora, which plays an important role in the health of the host. Many studies have also confirmed that the composition and function of the intestinal flora can be changed through the training chain. Changes in the composition of intestinal microbes can affect exercise performance, energy metabolism, oxidative stress, immune function, inflammation, and tissue repair. Therefore, maintaining a healthy gut microbial balance is essential for athletes' health, training, nutritional status, and athletic performance. This project intends to use metagenomics, proteomics, and metabolomics and other technologies to systematically explore the effects of different training periods and dietary interventions on the intestinal flora of muscle strength and endurance athletes. , Protein expression and the influence of metabolites. In the plan, explore the differences in the intestinal flora between muscle strength and endurance sports athletes during the preparation period, competition period, and transition period, and collect blood and feces to perform protein and metabolite molecular changes. It is hoped that through the smooth implementation of this research project, the research results can be applied to personalized diet planning, improve intestinal adaptability and the effectiveness of sports nutrition intervention, and then adjust athletes' status and improve sports performance to win the highest honor for the country in the arena.

ELIGIBILITY:
Inclusion Criteria:

* 20-30 years old healthy muscle strength and endurance sports athletes

Exclusion Criteria:

1. Exclude cardiovascular disease, hypertension, metabolic disease, asthma, or neuromuscular sports injuries within six months, etc.
2. Exclude those who regularly take lactic acid bacteria-related foods for a long time
3. Exclude students and related stakeholders under the guidance of the project host

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Recruitment of 12 healthy muscle and endurance athletes from the National Sports University
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-02-03 (Estimated); Study Completion 2021-02-03 (Estimated)

PRIMARY OUTCOMES:
Differences in intestinal flora of athletes in sports during preparation, competition and transition periods | 2021/1/1-2021/2/28
  asparate aminotransferase、alanine aminotransferase、albumin、blood urea nitrogen Creatinine、uric acid、total cholesterol、triacylglycerol、High-density lipoprotein、Low density lipoprotein、Free fatty acid、glucose、creatine kinase、gut microbiota

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Sport University, Taoyuan, Taiwan